CLINICAL TRIAL: NCT01087788
Title: Phase 3, Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Certolizumab Pegol in Subjects With Adult-Onset Active and Progressive Psoriatic Arthritis (PsA)
Brief Title: Certolizumab Pegol in Subjects With Adult Onset Active and Progressive Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PsA001; 2009-011720-59 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2017-01

CONDITIONS: Arthritis, Psoriatic
Keywords: Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- CZP 200 mg Q2W (Experimental): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
  At every visit, subjects received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
  Interventions: Biological: CZP 200 mg Q2W; Other: Placebo
- CZP 400 mg Q4W (Experimental): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 8 onwards.
  Subjects received 2 injections of Placebo every 4 weeks in between the 2 injections of 200 mg CZP to maintain the study blind.
  Interventions: Biological: CZP 400 mg Q4W; Other: Placebo
- Placebo (Placebo Comparator): Matching Placebo to Certolizumab Pegol (CZP) injections from Week 0 to Week 24. Placebo subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group and were re-randomized to either CZP 200 mg Q2W or CZP 400 mg Q4W arm on Week 16.
  After 24 weeks, all subjects were re-randomized to active treatment with CZP 200 mg every two weeks (Q2W) or CZP 400 mg every four weeks (Q4W).
  Interventions: Other: Placebo
- Placebo to CZP 200 mg escape on Week 16 (Other): Matching Placebo to CZP injections from Week 0 to Week 16. Subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16 and were treated with three loading doses of CZP 400 mg sc on Weeks 16, 18 and 20, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 22 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 200 mg Q2W; Other: Placebo
- Placebo to CZP 400 mg escape on Week 16 (Other): Matching Placebo to CZP injections from Week 0 to Week 16. Subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group on Week 16 and were treated with three loading doses of CZP 400 mg sc on Weeks 16, 18 and 20, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 24 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 400 mg Q4W; Other: Placebo
- Placebo to CZP 200 mg on Week 24 (Other): Matching Placebo to CZP injections from Week 0 to Week 24. Three loading doses of CZP 400 mg sc were given on Weeks 24, 26 and 28, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 30 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 200 mg Q2W; Other: Placebo
- Placebo to CZP 400 mg on Week 24 (Other): Matching Placebo to CZP injections from Week 0 to Week 24. Three loading doses of CZP 400 mg sc were given on Weeks 24, 26 and 28, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 32 onwards. Additionally, Placebo injections were administered as appropriate in order to maintain the study blind.
  Interventions: Biological: CZP 400 mg Q4W; Other: Placebo

INTERVENTIONS:
Biological: CZP 200 mg Q2W — 200 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 2 weeks (Q2W).
  Other Names: Cimzia; Certolizumab Pegol
  Arms: CZP 200 mg Q2W; Placebo to CZP 200 mg escape on Week 16; Placebo to CZP 200 mg on Week 24
Biological: CZP 400 mg Q4W — 400 mg subcutaneous (sc) injection of Certolizumab Pegol (CZP) every 4 weeks (Q4W).
  Other Names: Cimzia; Certolizumab Pegol
  Arms: CZP 400 mg Q4W; Placebo to CZP 400 mg escape on Week 16; Placebo to CZP 400 mg on Week 24
Other: Placebo — Matching Placebo to CZP injection.

SUMMARY:
Phase 3, multicenter, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy and safety of Certolizumab Pegol (CZP) in subjects with adult onset active and progressive Psoriatic Arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult-onset Psoriatic Arthritis (PsA) of at least 6 months' duration as defined by the Classification Criteria for Psoriatic Arthritis (CASPAR criteria)
* Active Psoriatic Skin Lesions or a documented history of Psoriasis
* Active Arthritis with ≥ 3 tender joints at Screening and Baseline, ≥ 3 swollen joints at Screening and Baseline and fulfilling at least 1 of the following 2 criteria during the Screening Period:

  1. Erythrocyte Sedimentation Rate (ESR) (Westergren) ≥ 28 mm/hour
  2. C-reactive protein (CRP) > Upper Limit Normal (ULN)
* Failure to 1 or more treatment with Disease-Modifying Anti-Rheumatic Drugs (DMARDs)

Exclusion Criteria:

* Diagnosis of any other inflammatory Arthritis or known diagnosis of Fibromyalgia
* Exposure to more than 1 Tumor Necrosis Factor α (TNFα) antagonist or to more than 2 previous biological response modifiers for PsA or Psoriasis
* Any non-biological systemic treatment of Psoriasis; phototherapy; topical agents
* History of chronic or recurrent infections
* High risk of infection
* Live vaccination within the 8 weeks prior to Baseline
* Concurrent malignancy or a history of malignancy
* Class III or IV congestive Heart Failure - New York Heart Association (NYHA)
* Demyelinating disease of the central nervous system
* Clinically significant laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 UCB
Locations (92):
- United States (27):
  - 961, Birmingham, Alabama
  - 953, Tuscaloosa, Alabama
  - 954, Peoria, Arizona
  - 971, Scottsdale, Arizona
  - 966, Palm Desert, California
  - 952, San Diego, California
  - 957, Aventura, Florida
  - 962, Fort Lauderdale, Florida
  - 959, Orange Park, Florida
  - 958, Vero Beach, Florida
  - 964, Hagerstown, Maryland
  - 960, Kalamazoo, Michigan
  - 969, Eagan, Minnesota
  - 984, Flowood, Mississippi
  - 965, Florissant, Missouri
  - 950, St Louis, Missouri
  - 985, Brooklyn, New York
  - 963, Asheville, North Carolina
  - 976, Cleveland, Ohio
  - 951, Middleburg Heights, Ohio
  - 970, Oklahoma City, Oklahoma
  - 982, Portland, Oregon
  - 972, Duncansville, Pennsylvania
  - 975, Dallas, Texas
  - 978, Houston, Texas
  - 967, San Antonio, Texas
  - 968, Seattle, Washington
- Argentina (8):
  - 700, Buenos Aires
  - 704, Buenos Aires
  - 707, Buenos Aires
  - 705, Córdoba
  - 706, Rosario
  - 710, San Juan
  - 702, San Miguel de Tucumán
  - 708, San Miguel de Tucumán
- Belgium (2):
  - 152, Ghent
  - 151, Liège
- Brazil (4):
  - 750, Curitiba
  - 757, Goiás
  - 761, Goiâna
  - 753, Porto Alegre
- Canada (5):
  - 907, Victoria, British Columbia
  - 900, St. John's, Newfoundland and Labrador
  - 904, Toronto, Ontario
  - 910, Windsor, Ontario
  - 905, Trois-Rivires, Quebec
- Czechia (6):
  - 504, Brno
  - 501, Hlučín
  - 500, Pardubice
  - 502, Prague
  - 505, Terezín
  - 503, Zlín
- France (3):
  - 206, Montpellier
  - 204, Paris
  - 202, Tours
- Germany (9):
  - 252, Bad Nauheim
  - 257, Berlin
  - 258, Berlin
  - 262, Frankfurt
  - 255, Freiburg im Breisgau
  - 254, Hamburg
  - 253, Leipzig
  - 263, München
  - 256, Ratingen
- Hungary (6):
  - 303, Budapest
  - 304, Budapest
  - 302, Debrecen
  - 301, Gyula
  - 306, Miskolc
  - 300, Veszprém
- 100, Dublin, Ireland
- Italy (2):
  - 352, Ancona
  - 350, Pisa
- Mexico (2):
  - 802, Cuernavaca
  - 803, Mexico City
- Poland (10):
  - 458, Bialystok
  - 452, Dąbrówka
  - 455, Elblag
  - 459, Gdansk
  - 457, Krakow
  - 450, Lublin
  - 454, Poznan
  - 453, Torun
  - 456, Warsaw
  - 462, Warsaw
- Spain (4):
  - 555, Madrid
  - 550, Mérida
  - 552, Santiago de Compostela
  - 553, Seville
- United Kingdom (3):
  - 605, Barnsley
  - 602, London
  - 601, Salford

REFERENCES:
- [Result] Mease PJ, Fleischmann R, Deodhar AA, Wollenhaupt J, Khraishi M, Kielar D, Woltering F, Stach C, Hoepken B, Arledge T, van der Heijde D. Effect of certolizumab pegol on signs and symptoms in patients with psoriatic arthritis: 24-week results of a Phase 3 double-blind randomised placebo-controlled study (RAPID-PsA). Ann Rheum Dis. 2014 Jan;73(1):48-55. doi: 10.1136/annrheumdis-2013-203696. Epub 2013 Aug 13. PMID 23942868
- [Result] van der Heijde D, Fleischmann R, Wollenhaupt J, Deodhar A, Kielar D, Woltering F, Stach C, Hoepken B, Arledge T, Mease PJ. Effect of different imputation approaches on the evaluation of radiographic progression in patients with psoriatic arthritis: results of the RAPID-PsA 24-week phase III double-blind randomised placebo-controlled study of certolizumab pegol. Ann Rheum Dis. 2014 Jan;73(1):233-7. doi: 10.1136/annrheumdis-2013-203697. Epub 2013 Aug 13. PMID 23942869
- [Result] van der Heijde D, Deodhar A, FitzGerald O, Fleischmann R, Gladman D, Gottlieb AB, Hoepken B, Bauer L, Irvin-Sellers O, Khraishi M, Peterson L, Turkiewicz A, Wollenhaupt J, Mease PJ. 4-year results from the RAPID-PsA phase 3 randomised placebo-controlled trial of certolizumab pegol in psoriatic arthritis. RMD Open. 2018 Mar 14;4(1):e000582. doi: 10.1136/rmdopen-2017-000582. eCollection 2018. PMID 29556416
- [Derived] Walsh JA, Gottlieb AB, Hoepken B, Nurminen T, Mease PJ. Efficacy of certolizumab pegol with and without concomitant use of disease-modifying anti-rheumatic drugs over 4 years in psoriatic arthritis patients: results from the RAPID-PsA randomized controlled trial. Clin Rheumatol. 2018 Dec;37(12):3285-3296. doi: 10.1007/s10067-018-4227-7. Epub 2018 Sep 6. PMID 30191421
- [Derived] van der Heijde D, Deodhar A, Fleischmann R, Mease PJ, Rudwaleit M, Nurminen T, Davies O. Early Disease Activity or Clinical Response as Predictors of Long-Term Outcomes With Certolizumab Pegol in Axial Spondyloarthritis or Psoriatic Arthritis. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1030-1039. doi: 10.1002/acr.23092. Epub 2017 Jun 2. PMID 27696727
- [Derived] Osterhaus JT, Purcaru O. Discriminant validity, responsiveness and reliability of the arthritis-specific Work Productivity Survey assessing workplace and household productivity in patients with psoriatic arthritis. Arthritis Res Ther. 2014 Jul 4;16(4):R140. doi: 10.1186/ar4602. PMID 24996416
- [Derived] Kavanaugh A, Gladman D, van der Heijde D, Purcaru O, Mease P. Improvements in productivity at paid work and within the household, and increased participation in daily activities after 24 weeks of certolizumab pegol treatment of patients with psoriatic arthritis: results of a phase 3 double-blind randomised placebo-controlled study. Ann Rheum Dis. 2015 Jan;74(1):44-51. doi: 10.1136/annrheumdis-2014-205198. Epub 2014 Jun 18. PMID 24942382
- [Derived] Gladman D, Fleischmann R, Coteur G, Woltering F, Mease PJ. Effect of certolizumab pegol on multiple facets of psoriatic arthritis as reported by patients: 24-week patient-reported outcome results of a phase III, multicenter study. Arthritis Care Res (Hoboken). 2014 Jul;66(7):1085-92. doi: 10.1002/acr.22256. PMID 24339179
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll patients in March 2010 and concluded in August 2015.
Pre-assignment Details: The study included a 24-week Double-Blind, a 24-week Dose-Blind, and an Open-Label Treatment Period.
  409 subjects are included in Randomized Set (RS) shown in the Participant Flow, which is an Intention- to- Treat (ITT) dataset.
Groups:
- Placebo: Matching Placebo (PBO) to Certolizumab Pegol (CZP) injections from Week 0 to Week 24. Placebo subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group and were re-randomized to either CZP 200 mg Q2W or CZP 400 mg Q4W arm on Week 16.
  After 24 weeks, all subjects were re-randomized to active treatment with CZP 200 mg every two weeks (Q2W) or CZP 400 mg every four weeks (Q4W).
Period: 24-weeks Double-blind Period
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W
Started | 136 | 138 | 135
Received CZP 200 mg Q2W at 16 Weeks | 30 (30 subjects left the Placebo group and were re-randomized to CZP 200 mg Q2W on Week 16.) | 0 (not applicable for this arm) | 0 (not applicable for this arm)
Received CZP 400 mg Q4W at 16 Weeks | 29 (29 subjects left the Placebo group and were re-randomized to CZP 400 mg Q4W on Week 16.) | 0 (not applicable for this arm) | 0 (not applicable for this arm)
Completed | 120 | 128 | 120
Not Completed | 16 | 10 | 15
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 2 | 5
Not completed — AE, serious fatal | 0 | 1 | 1
Not completed — AE, serious non-fatal | 0 | 2 | 3
Not completed — AE, non-serious non-fatal | 2 | 1 | 2
Not completed — AE, unknown type | 0 | 0 | 1
Not completed — Patient (P) does not want to attend | 1 | 0 | 0
Not completed — Protocol violation (decision of monitor) | 0 | 1 | 0
Not completed — Exclusion criteria were not met | 0 | 1 | 0
Not completed — P cannot comply with scheduled visits | 0 | 0 | 1
Period: 24-weeks Dose-blind Period
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W
Started | 120 | 128 | 120
Received CZP 200 mg Q2W at 24 Weeks | 60 (Sum of subjects re-randomized to CZP 200mg Q2W at week 16 (30 subjects) and at week 24 (30 subjects)) | 0 (not applicable for this arm) | 0 (not applicable for this arm)
Received CZP 400 mg Q2W at 24 Weeks | 60 (Sum of subjects re-randomized to CZP 400mg Q2W at week 16 (29 subjects) and at week 24 (31 subjects)) | 0 (not applicable for this arm) | 0 (not applicable for this arm)
Completed | 113 | 123 | 114
Not Completed | 7 | 5 | 6
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — AE, serious fatal | 0 | 1 | 0
Not completed — AE, serious non-fatal | 2 | 1 | 2
Not completed — AE, non-serious non-fatal | 2 | 1 | 1
Not completed — Sponsor decision following missed visits | 1 | 0 | 0
Not completed — Patient moved | 0 | 0 | 1
Period: Open-Label Period (OL-P)
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W
Started | 111 (2 subj. completed the Dose-Blind Period, then withdrew from the study rather than entering the OL-P.) | 121 (2 subj. completed the Dose-Blind Period, then withdrew from the study rather than entering the OL-P.) | 114
Completed | 81 | 97 | 86
Not Completed | 30 | 24 | 28
Not completed — Lack of Efficacy | 4 | 2 | 3
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 4 | 2
Not completed — Withdrawal by Subject | 13 | 8 | 10
Not completed — AE, serious fatal | 2 | 0 | 1
Not completed — AE, serious non-fatal | 1 | 3 | 4
Not completed — AE, non-serious non-fatal | 6 | 4 | 4
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 0 | 1 | 0
Not completed — AE, non-serious unknown | 1 | 0 | 0
Not completed — Sponsor request | 1 | 0 | 0
Not completed — Principal investigator decision | 0 | 1 | 2
Not completed — No participation in study extension | 0 | 0 | 1
Not completed — Personal reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 409 subjects are included in Randomized Set (RS) shown in Baseline Characteristics, which is an Intention-to-Treat (ITT) dataset.
Arm/Group | Placebo | CZP 200 mg Q2W | CZP 400 mg Q4W | Total Title
Number analyzed (Participants) | 136 | 138 | 135 | 409
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 129 | 126 | 128 | 383
  >=65 years | 7 | 12 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.1) | 48.2 (12.3) | 47.1 (10.8) | 47.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 74 | 73 | 226
  Male | 57 | 64 | 62 | 183

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20 (ACR20) Response at Week 12
Description: ACR20 responders are those subjects with at least 20 % improvement from Baseline (BL) for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS).
Time Frame: Week 12
Population: Intention-to-treat dataset was the Randomized Set (RS). RS with non-responder imputation: subjects who withdrew for any reason or placebo subjects who used escape medication are considered as nonresponders from drop out timepoint or when escape therapy was initiated. Subjects with missing data at a visit are non-responders for that visit, too.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo (Randomized Set): Matching Placebo to Certolizumab Pegol (CZP) injections from Week 0 to Week 24. Placebo subjects who did not achieve certain predefined response criteria at both Weeks 14 and 16 left the Placebo group and were re-randomized to either CZP 200 mg Q2W or CZP 400 mg Q4W arm on Week 16.
  After 24 weeks, all subjects were re-randomized to active treatment with CZP 200 mg every two weeks (Q2W) or CZP 400 mg every four weeks (Q4W).
- CZP 200 mg Q2W (Randomized Set): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
  At every visit, subjects received one injection of 200 mg CZP and one injection of Placebo to maintain the study blind.
- CZP 400 mg Q4W (Randomized Set): Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 400 mg CZP sc every 4 weeks (Q4W) from Week 8 onwards.
  Subjects received 2 injections of Placebo every 4 weeks in between the 2 injections of 200 mg CZP to maintain the study blind.
Arm/Group | Placebo (Randomized Set) | CZP 200 mg Q2W (Randomized Set) | CZP 400 mg Q4W (Randomized Set)
Number analyzed (Participants) | 136 | 138 | 135
percentage of participants | 24.3 [17.1 to 31.5] | 58.0 [49.7 to 66.2] | 51.9 [43.4 to 60.3]
Statistical Analysis 1: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W (Randomized Set); A hierarchical test procedure was applied to protect the overall significance level for the multiplicity of dose groups and endpoints. Conditional on the first test being significant, the second hypothesis was tested with the same alpha level of 5 %. Statistical testing for the following hypotheses was performed only if the previous null hypothesis in the hierarchy was rejected; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — Difference of Certolizumab Pegol 200 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using a standard two-sided Wald asymptotic test with a 5 % alpha level; Difference in Percentages = 33.7, 95% CI 2-sided [22.8 to 44.6]
Statistical Analysis 2: Comparison: Placebo (Randomized Set) vs CZP 400 mg Q4W (Randomized Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — Difference of Certolizumab Pegol 400 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using a standard two-sided Wald asymptotic test with a 5 % alpha level; Difference in Percentages = 27.6, 95% CI 2-sided [16.5 to 38.7]

2. Primary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) in Modification for Psoriatic Arthritis at Week 24
Description: Van der Heijde modified Total Sharp Score (mTSS) is a methodology to assess the degree of joint damage by quantifying the extent of bone erosions and joint space narrowing for 64 and 52 joints, respectively, with higher scores representing greater damage. mTSS (bone erosions) ranges from 0 (best possible outcome) to 320 (worst possible outcome); mTSS (joint space narrowing) ranges from 0 (best possible outcome) to 208 (worst possible outcome); and total score ranges from 0 (best possible outcome) to 528 (worst possible outcome). For the pre-defined analysis of this outcome measure, 0 was used for Baseline and the maximum observed mTSS value was used for Week 24 for those subjects which had less than 2 radiographs. The re-analysis is restricted to those subjects in the Randomized Set who have at least 2 x-ray values at scheduled visits, which are at least 8 weeks apart.
Time Frame: From Baseline to Week 24
Population: Intention-to-treat dataset was the Randomized Set (RS). RS with imputation: for subjects who withdrew for any reason, or subjects with missing Week 24 measurements, or placebo subjects who used escape medication, scores are linearly extrapolated from the last two radiographs prior to early withdrawal or Week 24 or before receiving CZP.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set): This combined group includes subjects of the two treatment arms CZP 200 mg Q2W and CZP 400 mg Q4W used in some analyses.
  Subjects received Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W)/ 400 mg CZP sc every 4 weeks (Q4W) from Week 6/ Week 8 onwards.
  Subjects in both CZP arms received additional placebo injections to maintain the study blind.
Arm/Group | Placebo (Randomized Set) | CZP 200 mg Q2W (Randomized Set) | CZP 400 mg Q4W (Randomized Set) | CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set)
Number analyzed (Participants) | 136 | 138 | 135 | 273
units on a scale
  Pre-defined results | 28.92 [13.73 to 44.11] | 11.52 [-3.40 to 26.45] | 25.05 [9.48 to 40.61] | 18.28 [6.34 to 30.23]
  Re-analysis results ( n = 123, 130, 123, 253) | 0.18 [0.04 to 0.33] | -0.02 [-0.16 to 0.11] | 0.09 [-0.05 to 0.23] | 0.03 [-0.08 to 0.14]
Statistical Analysis 1: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set); A hierarchical test procedure was applied to protect the overall significance level for the multiplicity of dose groups and endpoints. Conditional on the first test being significant, the second hypothesis was tested with the same alpha level of 5 %. Statistical testing for the following hypotheses was performed only if the previous null hypothesis in the hierarchy was rejected. This is the pre-defined primary analysis; Test type: Superiority or Other; p = 0.203, ANCOVA — Diff. of CZP 200mg+400mg versus PBO (and corresponding 95% Confidence Interval and p-value) were estimated using an ANCOVA model with treatment, region and prior Tumor Necrosis Factor(TNF)-antagonist exposure as factors & BL mTSS score as a covariate; Least Square Mean Difference (Net) = -10.64, 95% CI 2-sided [-27.05 to 5.77], Standard Error of Mean 8.35
Statistical Analysis 2: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W (Randomized Set); A hierarchical test procedure was applied to protect the overall significance level for the multiplicity of dose groups and endpoints.Conditional on the 1st test being significant, the 2nd hypothesis was tested with the same alpha level of 5%. Stat. testing for the following hypotheses was performed only if the previous null hypothesis in the hierarchy was rejected Re-analysis approach, restricted to subjects in the RS who have at least 2 x-ray values at scheduled visits (at least 8 wks apart); Test type: Superiority or Other; p = 0.017, ANCOVA — Difference of CZP 200 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using an ANCOVA model with treatment, region and prior TNF-antagonist exposure as factors and Baseline mTSS score as a covariate; Least Square Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.38 to -0.04], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Placebo (Randomized Set) vs CZP 400 mg Q4W (Randomized Set); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.261, ANCOVA — Difference of CZP 400 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using an ANCOVA model with treatment, region and prior TNF-antagonist exposure as factors and Baseline mTSS score as a covariate; Least Square Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.27 to 0.07], Standard Error of Mean 0.09

3. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at Week 24
Description: ACR20 responders are those subjects with at least 20 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGADA-VAS).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Randomized Set) | CZP 200 mg Q2W (Randomized Set) | CZP 400 mg Q4W (Randomized Set)
Number analyzed (Participants) | 136 | 138 | 135
percentage of participants | 23.5 [16.4 to 30.7] | 63.8 [55.7 to 71.8] | 56.3 [47.9 to 64.7]
Statistical Analysis 1: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W (Randomized Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — [p-value comment as in outcome 1, analysis 1]; Difference in Percentages = 40.2, 95% CI 2-sided [29.5 to 51.0]
Statistical Analysis 2: Comparison: Placebo (Randomized Set) vs CZP 400 mg Q4W (Randomized Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — [p-value comment as in outcome 1, analysis 2]; Difference in Percentages = 32.8, 95% CI 2-sided [21.8 to 43.8]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 24
Description: The HAQ-DI is a measure of function in Arthritis. There are 20 items in eight categories that represent a comprehensive set of functional activities on a scale from 0 (without difficulty) to 3 (unable to perform without assistance). The category scores are averaged into an overall HAQ-DI from 0 to 3. Scores of 0 to 1 generally represent mild to moderate difficulty, 1 to 2 represent moderate to severe disability, and 2 to 3 indicate severe to very severe disability. A negative value in HAQ-DI change from Baseline indicates an improvement from Baseline. The higher the negative value, the higher the improvement.
Time Frame: From Baseline to Week 24
Population: Intention-to-treat dataset was the Randomized Set (RS). RS with Last Observation Carried Forward (LOCF): for subjects who withdrew for any reason, or subjects with missing Week 24 measurements, or placebo subjects who used escape medication, last observation prior to early withdrawal or Week 24 or before receiving CZP is carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Randomized Set) | CZP 200 mg Q2W (Randomized Set) | CZP 400 mg Q4W (Randomized Set) | CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set)
Number analyzed (Participants) | 136 | 138 | 135 | 273
units on a scale | -0.19 [-0.29 to -0.09] | -0.54 [-0.64 to -0.44] | -0.46 [-0.56 to -0.36] | -0.50 [-0.58 to -0.42]
Statistical Analysis 1: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Difference of CZP 200 mg + 400 mg vs. Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using an ANCOVA model with treatment, region and prior TNF-antagonist exposure as factors and Baseline HAQ-DI score as a covariate; Least Square Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.42 to -0.20], Standard Error of Mean 0.06

5. Secondary Outcome: Psoriasis Area Severity Index (PASI75) Response at Week 24 in the Subgroup of Subjects With Psoriasis (PSO) Involving at Least 3 % Body Surface Area (BSA) at Baseline
Description: The PASI75 response assessments are based on at least 75 % improvement in the PASI score from Baseline. The PASI score is a measure of the average redness, thickness, and scaliness of the psoriatic skin lesions (each graded on a 0 to 4 scale), weighted by the area of involvement.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Randomized Set) | CZP 200 mg Q2W (Randomized Set) | CZP 400 mg Q4W (Randomized Set) | CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set)
Number analyzed (Participants) | 86 | 90 | 76 | 166
percentage of participants | 15.1 [7.5 to 22.7] | 62.2 [52.2 to 72.2] | 60.5 [49.5 to 71.5] | 61.4 [54.0 to 68.8]
Statistical Analysis 1: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wald-test, 2-sided — Difference of Certolizumab Pegol 200 mg + 400 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using a standard two-sided Wald asymptotic test with a 5 % alpha level; Difference in Percentages = 46.3, 95% CI 2-sided [35.7 to 56.9]

6. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 48
Description: Van der Heijde modified Total Sharp Score (mTSS) is a methodology to assess the degree of joint damage by quantifying the extent of bone erosions and joint space narrowing for 64 and 52 joints, respectively, with higher scores representing greater damage. mTSS (bone erosions) ranges from 0 (best possible outcome) to 320 (worst possible outcome); mTSS (joint space narrowing) ranges from 0 (best possible outcome) to 208 (worst possible outcome); and total score ranges from 0 (best possible outcome) to 528 (worst possible outcome).
  For the analysis of this outcome measure, the change from Baseline to Week 48 was imputed using the median change from Baseline among all subjects for those subjects, which had less than 2 radiographs. The post-hoc analysis presented here is based on the subgroup of subjects which had a Baseline mTSS value greater than 6.
Time Frame: From Baseline to Week 48
Population: Randomized Set (RS) with imputation: for subjects who withdrew for any reason, or subjects with missing Week 48 measurements, and for all placebo subjects after the switch to CZP, Week 48 scores are linearly extrapolated from the last two available radiographs prior to early withdrawal or Week 24 or before receiving CZP.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Randomized Set) | CZP 200 mg Q2W (Randomized Set) | CZP 400 mg Q4W (Randomized Set) | CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set)
Number analyzed (Participants) | 136 | 138 | 135 | 273
units on a scale
  Predefined results: Overall | 0.32 [0.10 to 0.55] | 0.15 [-0.07 to 0.37] | 0.11 [-0.12 to 0.34] | 0.13 [-0.05 to 0.31]
  Post-hoc results: Basel. mTSS > 6 (n=61,65,65,130) | 0.78 [0.31 to 1.25] | 0.31 [-0.15 to 0.77] | 0.22 [-0.24 to 0.67] | 0.26 [-0.09 to 0.62]
Statistical Analysis 1: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set); A hierarchical test procedure was applied to protect the overall significance level for the multiplicity of dose groups and endpoints. Conditional on the first test being significant, the second hypothesis was tested with the same alpha level of 5 %. Statistical testing for the following hypotheses was performed only if the previous null hypothesis in the hierarchy was rejected. This is the predefined analysis; Test type: Superiority or Other; p = 0.127, ANCOVA — Difference of CZP 200 mg + 400 mg versus Placebo (and corresponding 95 % Confidence Interval and p-value) were estimated using an ANCOVA model with treatment, region and prior TNF-antagonist exposure as factors and Baseline mTSS score as a covariate; Least Square Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.43 to 0.05], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo (Randomized Set) vs CZP 200 mg Q2W and CZP 400 mg Q4W (Randomized Set); A hierarchical test procedure was applied to protect the overall significance level for the multiplicity of dose groups and endpoints. Conditional on the first test being significant, the second hypothesis was tested with the same alpha level of 5 %. Statistical testing for the following hypotheses was performed only if the previous null hypothesis in the hierarchy was rejected. This is the post-hoc analysis for the subgroup 'Baseline mTSS > 6'; Test type: Superiority or Other; p = 0.048, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Square Mean Difference (Net) = -0.52, 95% CI 2-sided [-1.04 to -0.01], Standard Error of Mean 0.26

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Baseline (Week 0) over the whole Double-Blind, Dose-Blind and Open-Label Period up to Week 216.
Description: As per study design, placebo (PBO) arm subjects shifted either at Week (Wk) 16 or 24 to CZP treatment. Thus, PBO arm had lower exposure compared to the CZP arms. The exposure imbalance across treatment arms could lead to misinterpretation & questionable conclusions comparing simple counts & percentages of AEs. Thus, AEs reported while the patient was on PBO-treatment are not included.
Groups:
- All CZP 200 mg Q2W: This arm includes all subjects who were randomized to CZP 200 mg Q2W at Baseline and those subjects who escaped or were re-randomized from Placebo to CZP 200 mg Q2W.
  Subjects received one injection of 200 mg CZP and one injection of Placebo every two weeks to maintain the study blind.
- All CZP 400 mg Q4W: This arm includes all subjects who were randomized to CZP 400 mg Q4W at Baseline and those subjects who escaped or were re-randomized from Placebo to CZP 400 mg Q4W.
  Subjects received two injections of Placebo every four weeks in between the two injections of 200 mg CZP to maintain the study blind.
- All CZP 200 mg + 400 mg: This arm shows all patients treated with Certolizumab Pegol (CZP) at least once. Hence, this arm is a combination of arm All CZP 200 mg Q2W and arm All CZP 400 mg Q4W.
Arm/Group | All CZP 200 mg Q2W | All CZP 400 mg Q4W | All CZP 200 mg + 400 mg
Serious Adverse Events (participants affected / at risk) | 49/198 | 51/195 | 100/393
Other Adverse Events (participants affected / at risk) | 158/198 | 153/195 | 311/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All CZP 200 mg Q2W (N=198) | All CZP 400 mg Q4W (N=195) | All CZP 200 mg + 400 mg (N=393)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (2)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (4) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pyoderma streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (7) | 8 (12)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 3 (3)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (2)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dysgraphia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Formication (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2)
Vulvar dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 4 (5)
Pregnancy of partner (Social circumstances) | 0 (0) | 1 (1) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All CZP 200 mg Q2W (N=198) | All CZP 400 mg Q4W (N=195) | All CZP 200 mg + 400 mg (N=393)
Diarrhoea (Gastrointestinal disorders) | 15 (20) | 11 (15) | 26 (35)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 9 (10) | 21 (23)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16) | 5 (9) | 19 (25)
Nausea (Gastrointestinal disorders) | 10 (11) | 8 (9) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 44 (81) | 49 (73) | 93 (154)
Nasopharyngitis (Infections and infestations) | 45 (87) | 42 (91) | 87 (178)
Pharyngitis (Infections and infestations) | 24 (44) | 27 (37) | 51 (81)
Bronchitis (Infections and infestations) | 28 (36) | 22 (29) | 50 (65)
Urinary tract infection (Infections and infestations) | 13 (18) | 26 (35) | 39 (53)
Sinusitis (Infections and infestations) | 19 (32) | 13 (33) | 32 (65)
Gastroenteritis (Infections and infestations) | 14 (18) | 8 (8) | 22 (26)
Oral herpes (Infections and infestations) | 10 (25) | 11 (18) | 21 (43)
Influenza (Infections and infestations) | 13 (15) | 8 (9) | 21 (24)
Tonsillitis (Infections and infestations) | 11 (11) | 8 (12) | 19 (23)
Rhinitis (Infections and infestations) | 10 (11) | 9 (9) | 19 (20)
Latent tuberculosis (Infections and infestations) | 6 (6) | 12 (12) | 18 (18)
Viral infection (Infections and infestations) | 9 (12) | 7 (7) | 16 (19)
Contusion (Injury, poisoning and procedural complications) | 15 (21) | 9 (10) | 24 (31)
Alanine aminotransferase increased (Investigations) | 17 (23) | 15 (25) | 32 (48)
Blood creatine phosphokinase increased (Investigations) | 15 (28) | 13 (25) | 28 (53)
Aspartate aminotransferase increased (Investigations) | 9 (13) | 11 (17) | 20 (30)
Gamma-glutamyltransferase increased (Investigations) | 8 (11) | 12 (15) | 20 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (28) | 22 (26) | 46 (54)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 24 (41) | 15 (23) | 39 (64)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (28) | 18 (28) | 38 (56)
Headache (Nervous system disorders) | 18 (19) | 17 (20) | 35 (39)
Dizziness (Nervous system disorders) | 5 (5) | 10 (10) | 15 (15)
Depression (Psychiatric disorders) | 11 (12) | 9 (12) | 20 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 14 (14) | 22 (23)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (13) | 16 (19)
Psoriasis (Skin and subcutaneous tissue disorders) | 22 (31) | 19 (21) | 41 (52)
Rash (Skin and subcutaneous tissue disorders) | 10 (16) | 9 (9) | 19 (25)
Hypertension (Vascular disorders) | 30 (33) | 16 (20) | 46 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days